CLINICAL TRIAL: NCT06376292
Title: A Prospective Single Arm Phase II Exploratory Study on the Combination of Whole Brain Radiotherapy and Thiotepa Intrathecal Injection for Systemic Treatment of Primary Diseases in the Treatment of Solid Tumor Leptomeningeal Metastasis
Brief Title: A Prospective Single Arm Phase II Exploratory Study on the Combination of Whole Brain Radiotherapy, Thiotepa Intrathecal Injection and Systemic Treatment of Primary Diseases in the Treatment of Solid Tumor Leptomeningeal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y2024-0106
Record Dates: First submitted 2024-02-27; First posted 2024-04-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Leptomeningeal Metastasis

STUDY DESIGN:
Intervention Model Description: Participants will receive a comprehensive treatment plan consisting mainly of HA-WBRT combined with intrathecal injection of Thiotepa. All eligible patients received intrathecal injection of Thiotepa twice a week for 1 week as induction treatment for 3 weeks, followed by once every week as consolidation therapy for 6 week and then once monthly as maintenance therapy, until progressive disease was observed or intolerance or adverse events (AEs) developed. The injection was administered by qualified individuals (certified personnel in the radiotherapy department of our hospital) . Thiotepa was injected 10mg each time, mixed with cerebrospinal fluid, and then injected slowly for 5-10 minutes. Evaluate the efficacy and safety every 6 cycles according to RANO-LM criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): Participants will receive a comprehensive treatment plan consisting mainly of whole brain 30Gy/10F radiotherapy combined with intrathecal injection of Thiotepa twice a week for a total of 4 weeks.
  Interventions: Drug: Intrathecal Injection of Thiotepa+Radiation+Systemic Treatment of Primary Diseases

INTERVENTIONS:
Drug: Intrathecal Injection of Thiotepa+Radiation+Systemic Treatment of Primary Diseases — Participants will receive a comprehensive treatment plan consisting mainly of whole brain 30Gy/10F radiotherapy combined with intrathecal injection of Thiotepa. The injection was administered by qualified individuals (certified personnel in the radiotherapy department of our hospital) twice a week for a total of 4 weeks. Thiotepa was injected 10mg each time, mixed with cerebrospinal fluid, and then injected slowly for 5-10 minutes.

SUMMARY:
The goal of this prospective, single-arm exploratory clinical study is to explore the safty and efficacy of whole-brain radiotherapy combined with Thiotepa intrathecal injection combined with systemic therapy for the primary disease in the treatment of leptoeningeal metastases in solid tumors

How works well was the combined therapy？ How safe was combined therapy？ Participants will continue systemic treatment, receive HA-WBRT combined with intrathecal injection of Thiotepa. Evaluate the efficacy and safety every 6 cycles.

Researchers will evaluate whether this combination treatment is safe and whether it is more effective than previous studies.

DETAILED DESCRIPTION:
Participants will receive a comprehensive treatment plan consisting mainly of HA-WBRT combined with intrathecal injection of Thiotepa. All eligible patients received intrathecal injection of Thiotepa twice a week for 1 week as induction treatment for 3 weeks, followed by once every week as consolidation therapy for 6 week and then once monthly as maintenance therapy, until progressive disease was observed or intolerance or adverse events (AEs) developed. The injection was administered by qualified individuals (certified personnel in the radiotherapy department of our hospital) . Thiotepa was injected 10mg each time, mixed with cerebrospinal fluid, and then injected slowly for 5-10 minutes. Evaluate the efficacy and safety every 6 cycles according to RANO-LM criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1) Voluntary participation in clinical research: fully understand and be informed of this study, and sign an informed consent form in writing; Willing to follow and capable of completing all experimental procedures.

  2) Age: ≥ 18 years old, both male and female. 3) Solid tumor patients diagnosed with meningeal metastasis according to the EANO-ESMO guidelines 4) Whole brain 6MX X-ray PTV D95/30Gy/10F regimen radiotherapy has been performed 5) CNS IPI ≥ 4. 6) An increase in serum LDH or involvement of more than one extranodal site. 7) ECOG score ≤ 2. 8) Expected survival time is at least 3 months. 9) Adequate organ and bone marrow function, without severe hematopoietic dysfunction, heart, lung, liver, kidney dysfunction, and immune deficiency (no blood transfusion, granulocyte colony-stimulating factor, or other related medical support received within 14 days prior to the use of the study drug):
  1. Blood routine: Absolute neutrophil count (ANC) ≥ 1.5'109/L (1500/mm3), platelet count ≥ 75'109/L, hemoglobin count ≥ 9 g/dL (if bone marrow is involved, platelet count ≥ 50'109/L, ANC ≥ 1.0'109/L, hemoglobin count ≥ 8 g/dL).
  2. Liver function: Serum bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 times the upper limit of normal value (if liver involvement occurs, AST is allowed, ALT ≤ 5 times the upper limit of normal value).
  3. Renal function: Serum creatinine ≤ 1.5 times the upper limit of normal value.
  4. Coagulation function: INR ≤ 1.5 times the upper limit of normal value; PT and APTT ≤ 1.5 times the upper limit of normal values (unless the subject is receiving anticoagulant treatment and PT and APTT are within the expected range of anticoagulant treatment during screening).

     10) Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.

     11) The serum pregnancy test is negative, and effective contraceptive measures are taken within 6 months from the signing of the informed consent form until the use of the last chemotherapy.

     12) Thyroid stimulating hormone (TSH), free thyroxine (FT4), or free triiodothyronine (FT3) are all within the normal range of ± 10%.

     13) Ophthalmic examination: including dilated pupil fundus examination, slit lamp examination, and fundus color photography.

     Exclusion Criteria:
* 1) Participating in other clinical studies, or the first study drug administration is less than 4 weeks after the end of the previous clinical study treatment.

  2) Has suffered from other malignant tumors within the past 5 years. 3) Patients who have received CNS guided treatment and prevention. 4) Patients with a known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.

  5) Patients with active autoimmune diseases or a history of hematological autoimmune diseases with a high risk of recurrence, including but not limited to immune related neuropathy, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain's syndrome, myasthenia gravis, systemic lupus erythematosus, connective tissue disease, scleroderma, inflammatory bowel cancer (including Crohn's disease and ulcerative colitis), autoimmune hepatitis Toxic epidermal necrolysis or Stevens Johnson syndrome.

  6) Patients with active chronic hepatitis B or active hepatitis C. Patients with positive hepatitis B B surface antigen or hepatitis C virus antibody in screening period must further pass the hepatitis B virus DNA drop test (not more than 1000 iu/ml) and HCV RNA test (not more than the lower limit of the test method), and can be included in the test only after the active hepatitis B or hepatitis C infection requiring treatment is excluded. Hepatitis B virus carriers, hepatitis B patients who are stable after drug treatment and cured hepatitis C patients can be included in the group.

  7) Suffer from active pulmonary tuberculosis. 8) Currently, there is interstitial lung disease or infectious pneumonia. 9) Active infections that require systematic anti infective treatment, including but not limited to bacterial, fungal, or viral infections.

  10) Screening for heart failure classified as Grade III or IV according to the New York Heart Association (NYHA) functional classification within the first 6 months, unstable angina, severe uncontrolled ventricular arrhythmias, and electrocardiograms showing acute ischemia or myocardial infarction.

  11) QTcF interval>480msec, unless secondary to bundle branch block. 12) Suffering from uncontrollable comorbidities, including but not limited to uncontrollable hypertension, active peptic ulcers, or hemorrhagic diseases.

  13) Individuals with a history of mental illness; Individuals with no or limited capacity for behavior.

  14) According to the researchers, the patient's underlying condition may increase their risk of receiving treatment with the investigational drug, or may cause confusion regarding the occurrence of toxic reactions and their judgment.

  15) Other researchers believe that patients who are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  The primary safety analysis will be conducted based on subjects who experience toxicity (as defined by CTCAE standards). CTCAE version 5.0 will be used to evaluate safety through reported adverse events.

SECONDARY OUTCOMES:
OS | 2 years
  overall survival
PFS | 2 years
  progression free survival
3-month OS | 3 months
  3-month overall survival
6-month OS | 6 months
  6-month overall survival
9-month OS | 9 months
  9-month overall survival
12-month OS | 12 months
  12-month overall survival
The disease control rate(DCR) | 2 years
  the proportion of patients who, according to internationally recognized criteria for alleviating evaluation, achieve response and stable disease (SD) after treatment and can maintain for the minimum duration requirement.
The objective response rate (ORR) | 2 years
  The sum of the proportion of responsive patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT06376292/Prot_002.pdf
  • Informed Consent Form (2024-01-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT06376292/ICF_003.pdf